CLINICAL TRIAL: NCT06558214
Title: OPTIMUS PRIME: Safety and Feasibility of OPTune GIO® Integrated With MRI-gUided Laser Ablation Surgery and Pembrolizumab for Recurrent GlIoblastoMa, A randomizEd Trial
Acronym: OPTIMUS PRIME
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB202400948; OCR45231 (Other: University of Florida)
Record Dates: First submitted 2024-08-14; First posted 2024-08-16 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Recurrent Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1: Optune GIO® pre-MLA; MLA; followed by Optune GIO® + Pembrolizumab post MLA (Experimental): Patients randomized to treatment arm 1 will start treatment with Optune GIO® for 3-7 days and undergo MLA and biopsy for tumor diagnosis and immune monitoring. Treatment with Optune GIO® will be paused prior to the MLA procedure until at least 10 days post MLA. Patients will then resume treatment with Optune GIO® and receive pembrolizumab 200 mg IV every 3 weeks (+/- 4 days) starting no sooner than 1 week after the start of Optune GIO®.
  Interventions: Drug: Pembrolizumab; Device: Optune GIO®; Device: NeuroBlate®
- Arm 2: Optune GIO®+Pembrolizumab pre-MLA; MLA; followed by Optune GIO® + Pembrolizumab post MLA (Experimental): Patients randomized to treatment arm 2, will start treatment with Optune GIO® for 3-10 days and receive one infusion of pembrolizumab before undergoing MLA/biopsy. Patients will resume Optune GIO® no earlier than 10 days post-surgery and receive pembrolizumab 200 mg IV every 3 weeks (+/- 4 days) starting no sooner than 1 week after the start of Optune GIO®.
  Interventions: Drug: Pembrolizumab; Device: Optune GIO®; Device: NeuroBlate®

INTERVENTIONS:
Drug: Pembrolizumab — Keytruda® is the trade name for pembrolizumab, which will be given as 200mg IV Q3 weeks. This treatment will continue for up to two years.
  Other Names: Keytruda
Device: Optune GIO® — .
  . Optune GIO® TTFields treatment will begin 3-7 days prior to MLA for Arm1 and 3-10 days prior to MLA for Arm 2.
  Other Names: TTFields
Device: NeuroBlate® — Treatment with NeuroBlate will occur one time at the beginning of the study.
  Other Names: MLA; LITT

SUMMARY:
In this study we are evaluating the safety and feasibility of the triple combination (TTFields, MLA, pembrolizumab) in adult patients diagnosed with recurrent or progressive glioblastoma (GBM) WHO Grade IV, IDH wild type or recurrent or progressive astrocytoma WHO grade IV.

DETAILED DESCRIPTION:
Twenty patients diagnosed with recurrent or progressive glioblastoma will be enrolled in this pilot study of safety and feasibility and receive the triple combination of Optune GIO®, MLA and pembrolizumab.

Patients will be identified and enrolled prior to initiation of treatment for recurrence and be randomized (1:1) to (each arm has 10 patients):

Arm 1: Optune GIO® pre-MLA; MLA; followed by Optune GIO® + Pembrolizumab post MLA

Arm 2: Optune GIO®+Pembrolizumab pre-MLA; MLA; followed by Optune GIO® + Pembrolizumab post MLA

Surgical resection/debulking is per standard of care and optional for the purpose of this study. The performing neurosurgeon will determine whether each patient will undergo surgery. For patients who undergo debulking surgery, MLA is expected to occur between 3-6 weeks post-surgery, when the performing surgeon assesses the procedure is safe.

Patients randomized to treatment arm 1 will start treatment with Optune GIO® for 3-7 days and undergo MLA and biopsy for tumor diagnosis and immune monitoring. Treatment with Optune GIO® will be paused prior to the MLA procedure until at least 10 days post MLA. Patients will then resume treatment with Optune GIO® and receive pembrolizumab 200 mg IV every 3 weeks (+/- 4 days) starting no sooner than 1 week after the start of Optune GIO®.

Patients randomized to treatment arm 2, will start treatment with Optune GIO® for 3-10 days and receive one infusion of pembrolizumab before undergoing MLA/biopsy. Patients will resume Optune GIO® no earlier than 10 days post-surgery and receive pembrolizumab 200 mg IV every 3 weeks (+/- 4 days) starting no sooner than 1 week after the start of Optune GIO®, Post MLA, patients may continue treatment with Optune GIO® and pembrolizumab for up to 2 years, or until disease progression, intolerable toxicity, whichever comes first.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years of age.
2. Diagnosis of recurrent or progressive glioblastoma, WHO Grade IV, IDH wild-Type or astrocytoma WHO grade IV.
3. Unequivocal evidence of tumor progression by brain MRI scan per RANO criteria. Patients who experience a second disease progression are eligible provided that they have not been previously treated with anti-angiogenic agents including bevacizumab (at the exception of bevacizumab radiation necrotic protocol)
4. A diagnostic contrast-enhanced MRI of the brain must be performed preoperatively, within 28 days prior to study enrollment.
5. There must be an interval of at least 12 weeks from the completion of radiation therapy to study registration unless there is unequivocal evidence for tumor recurrence per RANO criteria. When the interval is less than 12 weeks but more than 4 weeks from the completion of radiotherapy, the use of perfusion imaging and/or PET scan is allowed to differentiate between unequivocal evidence of tumor recurrence and pseudoprogression.
6. Karnofsky performance status (KPS) ≥60%.
7. Candidate for MLA based on the size, location, and shape of the recurrent tumor as determined by the performing neurosurgeon. Surgical resection/debulking prior to MLA is allowed per standard of care but is not required.
8. Candidate for Optune GIO® therapy.
9. Candidate for pembrolizumab.
10. Adequate bone marrow and organ function as defined below:

    1. ANC ≥ 1,500/mcL
    2. Platelets ≥ 100,000/mcL
    3. Hemoglobin ≥ 9 g/dL or ≥ 5.6 mmol/L (transfusion is allowed)
    4. Serum creatinine ≤ 1.5 x IULN OR creatinine clearance by Cockcroft-Gault ≥ 60 mL/min for patients with serum creatinine > 1.5 x IULN
    5. Serum total bilirubin ≤ 1.5 x IULN OR direct bilirubin ≤ IULN for patients with total bilirubin > 1.5 x IULN
    6. AST (SGOT) ≤ 3 x IULN
    7. ALT (SGPT) ≤ 3 x IULN
11. Participants of childbearing age must use effective contraception:

    Women of childbearing potential (WOCBP) must be using a highly effective method of contraception to avoid pregnancy throughout the study and for at least 24 weeks after the last dose of study drug to minimize the risk of pregnancy. Prior to study enrollment, women of childbearing potential must be advised of the importance of avoiding pregnancy during trial participation and the potential risk factors for an unintentional pregnancy.
    1. WOCBP include any woman who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation or oophorectomy) or who is not post-menopausal. Post-menopause is defined as:

       * Amenorrhea that has lasted for ≥ 12 consecutive months without another cause, or
       * For women with irregular menstrual periods who are taking hormone replacement therapy (HRT), a documented serum follicle-stimulating hormone (FSH) level of greater than 35 mIU/mL.
    2. Males with female partners of childbearing potential must agree to use physician-approved contraceptive methods (e.g., abstinence, condoms, vasectomy) throughout the study and should avoid conceiving children for 24 weeks following the last dose of study drug.
12. Ability of the patient to understand and willingness to sign an IRB approved written informed consent document

Exclusion Criteria:

1. Prior treatment with any anti-angiogenic agent, including bevacizumab.
2. Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
3. Prior treatment with a monoclonal antibody within 4 weeks prior to the projected first dose of pembrolizumab or has not recovered (i.e. ≤ grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
4. Prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to the projected first dose of pembrolizumab or has not recovered (i.e. ≤ grade 1 or at baseline) from adverse events due to a previously administered agent.

   Note: patients with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study.
5. Presence of infratentorial lesions, brainstem lesions, or lesions that are less than 5 mm from the hypophysis or cranial nerves.
6. Multifocal gliomas that are bilateral. Patients with unilateral multifocal gliomas may be eligible if their multifocal disease can be treated effectively and safely in a single MLA procedure. Also note that corpus callosal tumors are eligible even if they are bilateral as long as they satisfy the size and shape limits of MLA as determined by the performing neurosurgeon.
7. Presence of leptomeningeal metastases beyond the cranial vault. (Focal leptomeningeal enhancement allowable at the discretion of the principal investigator).
8. Requires corticosteroids equivalent to > 4mg dexamethasone daily.
9. Recent (within 8 weeks) history of CNS hemorrhage unless the hemorrhage is located within the tumor that will be removed en total during surgical debulking or ablated during MLA.
10. Requires therapeutic doses of anticoagulants unless anticoagulation can be safely discontinued per standard practice (e.g. first DVT for which anticoagulation has been at least 3 months and repeat imaging demonstrates resolution of DVT) or an IVC filter can be used in place of anticoagulation.
11. Received prior local therapy (stereotactic radiosurgery, brachytherapy, or carmustine wafers) to the proposed area of MLA treatment.
12. Received a live vaccine within 30 days prior to the projected initiation of study treatment (Optune GIO® for Arm 1 and LITT for Arm 2).
13. Currently receiving any other investigational agents or has participated in a study of an investigational agent or using an investigational device within 3 weeks of the projected initiation of study treatment (Optune GIO® for Arm 1 and LITT for Arm 2).
14. Has a diagnosis of immunodeficiency or is receiving any form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment (with the exception of daily dexamethasone ≤ 4 mg).
15. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
16. History of active autoimmune disease requiring systemic treatment within the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.

    (Note that prior autoimmune diseases at Grade 1 or 2 per CTCAE v. 4.0 in the last 2 years that were deemed related to prior use of immunotherapy, will be allowed under this protocol, provided that continuation or subsequent resumption of immunotherapy, regardless of whether systemic treatment had been given, did not result in worsening of signs and symptoms of the aforementioned autoimmune diseases)
17. History of (non-infectious) pneumonitis within the past 3 years that required steroids or current pneumonitis.

    (Note that patients with a history of pneumonitis in the past 3 years that was not aggravated by immunotherapy or that has clinically resolved or improved and has not recurred or progressed clinically with subsequent immunotherapy are eligible to participate in the study).
18. Pregnant and/or breastfeeding. Patient must have a negative serum or urine pregnancy test within 72 hours of study entry.
19. Known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected) infection.
20. Known history of active TB (bacillus tuberculosis).
21. Known history of HIV (HIV 1/2 antibodies).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants experiencing a DLT after receiving the triple combination (TTFields, MLA, pembrolizumab) in adult patients diagnosed with recurrent glioblastoma from both arms | baseline up to 3 months
  Patients who receive the combinatorial regimen will get the ongoing safety assessment with DLT </= 33% treated subjects
Percentage of participants treated with the triple combination (TTFields, MLA, pembrolizumab) in adult patients diagnosed with recurrent glioblastoma from both arms | baseline up to 3 months
  Feasibility is defined as the ability to successfully deliver the combinatorial treatment of MLA, optune GIO® and pembrolizumab to at least 67% of enrolled subjects who undergo MLA.

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Ghiaseddin, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Shands Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided